CLINICAL TRIAL: NCT03933306
Title: Impact of Intraoperative Goal-directed Blood Pressure Management and Dexmedetomidine on Outcomes of High-risk Patients After Major Abdominal Surgeries: a 2×2 Factorial Randomized Controlled Trial
Brief Title: Intraoperative Goal-directed Blood Pressure and Dexmedetomidine on Outcomes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anaesthesiology and Critical Care Medicine, Peking University First Hospital
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 2019-73
Record Dates: First submitted 2019-04-27; First posted 2019-05-01 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Blood Pressure; Dexmedetomidine; High-risk Patients; Abdominal Surgery; Postoperative Complications
Keywords: blood pressure management; dexmedetomidine; high-risk patients; abdominal surgery; postoperative organ injury
MeSH Terms: conditions — Postoperative Complications | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Intervention Model Description: This is a 2x2 factorial trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: For dexmedetomidine infusion, all the participants, care providers, investigators, outcomes assessors are masked. For blood pressure management, care providers, namely anesthesiologists, are not masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo+routine blood pressure management (Placebo Comparator): Placebo (normal saline) is administered during anesthesia. Blood pressure is managed according to routine practice.
  Interventions: Drug: Placebo; Other: Routine blood pressure management
- Dexmedetomidine+routine blood pressure management (Experimental): Dexmedetomidine is administered during anesthesia (0.6 mcg/kg for 10 min, then 0.5 mcg/kg/h). Blood pressure is managed according to routine practice.
  Interventions: Drug: Dexmedetomidine; Other: Routine blood pressure management
- Placebo+goal-directed blood pressure management (Experimental): Placebo (normal saline) is administered during anesthesia. Blood pressure is maintained within ±10% of baseline with noradrenaline infusion and fluid management.
  Interventions: Drug: Placebo; Other: Goal-directed blood pressure management
- Dexmedetomidine+goal-directed blood pressure management (Experimental): Dexmedetomidine is administered during anesthesia (0.6 mcg/kg for 10 min, then 0.5 mcg/kg/h). Blood pressure is maintained within ±10% of baseline with noradrenaline infusion and fluid management.
  Interventions: Drug: Dexmedetomidine; Other: Goal-directed blood pressure management

INTERVENTIONS:
Drug: Dexmedetomidine — Loading dose dexmedetomidine (0.6 mcg/kg for 10 min) administered before anesthesia induction, followed by a continuous infusion (0.5 mcg/kg/h) until 1 hour before the end of surgery.
  Other Names: Dexmedetomidine hydrochloride injection
  Arms: Dexmedetomidine+goal-directed blood pressure management; Dexmedetomidine+routine blood pressure management
Drug: Placebo — Loading dose placebo administered before anesthesia induction, followed by a continuous infusion until 1 hour before the end of surgery.
  Other Names: Normal saline
  Arms: Placebo+goal-directed blood pressure management; Placebo+routine blood pressure management
Other: Goal-directed blood pressure management — Blood pressure is maintained within ±10% of baseline with noradrenaline infusion and fluid management.
  Arms: Dexmedetomidine+goal-directed blood pressure management; Placebo+goal-directed blood pressure management
Other: Routine blood pressure management — Blood pressure is maintained according to routine practice, i.e., systolic blood pressure > 90 mmHg or within ±30% of baseline within intermittent ephedrine or phenylephrine.
  Arms: Dexmedetomidine+routine blood pressure management; Placebo+routine blood pressure management

SUMMARY:
Perioperative organ injuriy remain an important threat to patients undergoing major surgeries. Intraoperative hypotension is associated with an increase in postoperative morbidity and mortality. Whereas individualized intraoperative blood pressure management is likely to decrease the incidence of postoperative organ injury when compared with standard blood pressure management strategy. Dexmedetomidine, a highly selective alpha2 adrenergic agonist, has been shown to provide organ protective effects. This study aims to investigate the impact of intraoperative goal-directed blood pressure management and dexmedetomidine infusion on incidence of postoperative organ injury in high-risk patients undergoing major surgery.

DETAILED DESCRIPTION:
The number of patients undergoing surgeries is increasing worldwide. However, some patients develop complications or even die after surgery. Perioperative organ injury is the leading cause of the unfavorable outcomes.

Hypotension is not uncommon during major surgery and is highly responsible for the inadequate perfusion and organ injury. A recent study showed that individualized blood pressure management decreases the incidence of postoperative organ injury when compared with standard blood pressure management strategy.

Dexmedetomidine is a highly selective alpha2 adrenergic agonist. Previous studies showed that dexmedetomidine provides organ protection in various conditions. In a recent meta-analysis, perioperative dexmedetomidine reduceds the occurrence of postoperative delirium. However, whether it can reduce postoperative complications remains inconclusive.

This study aims to investigate the impact of intraoperative goal-directed blood pressure management and dexmedetomidine infusion on the incidence of postoperative organ injury in high-risk patients undergoing major abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 years or older;
* Scheduled to undergo abdominal surgery under general anesthesia with an expected duration of 2 hours or longer;
* With a preoperative acute kidney injury risk index of class III or higher (meet 4 or more of the following factors: age ≥56 years, male sex, active congestive heart failure, ascites, hypertension, emergency surgery, intraperitoneal surgery, mild or moderate renal insuffificiency, diabetes mellitus requiring oral or insulin therapy).

Exclusion Criteria:

* Severe uncontrolled hypertension (SBP>180 mmHg or diastolic blood pressure >110 mmHg);
* Acute or decompensated heart failure, acute coronary syndrome, or stroke within 1 month;
* Severe bradycardia (heart rate < 50 bpm), sick sinus syndrome, second-degree or higher atrioventricular block without pacemaker, atrial fibrillation, or frequent premature beats;
* Severe hepatic dysfunction (Child-Pugh C) or chronic kidney disease (glomerular filtration rate <30 ml/min/1.73 m2 or dependent on renal replacement therapy) ;
* Pregnant;
* Receiving dexmedetomidine or norepinephrine infusion before surgery;
* Do not provide written informed consent.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 496 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2020-10-29 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Incidence of organ injury and other complications within 30 days after surgery. | Up to 30 days after surgery.
  A composite endpoint including delirium, acute kidney injury, myocardial injury, and other complications after surgery.

SECONDARY OUTCOMES:
Incidence of organ injury and other complications within 7 days after surgery. | Up to 7 days after surgery.
  A composite endpoint including delirium, acute kidney injury, myocardial injury, and other complications after surgery.
Length of stay in the intensive care unit after surgery. | Up to 30 days after surgery.
  Length of stay in the intensive care unit after surgery.
Length of stay in hospital after surgery. | Up to 30 days after surgery.
  Length of stay in hospital after surgery.
30-day all-cause mortality. | Up to 30 days after surgery.
  Rate of death due to any cause within 30 days after surgery.
Overall survival after surgery. | Up to 3 years after surgery.
  Overall survival after surgery.
Disease-free survival after surgery. | Up to 3 years after surgery.
  Disease-free survival after surgery.
Quality of life of 3-year survivors: WHOQOL-BREF | At the end of 3 years after surgery.
  Quality of life is assessed with with the World Health Organization quality of life scale brief version (WHOQOL-BREF).
Cognition function of 3-year survivors. | At the end of 3 years after surgery.
  Cognitive function is assessed with the Telephone Interview for Cognitive Status-Modified (TICS-m).

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weiser TG, Haynes AB, Molina G, Lipsitz SR, Esquivel MM, Uribe-Leitz T, Fu R, Azad T, Chao TE, Berry WR, Gawande AA. Estimate of the global volume of surgery in 2012: an assessment supporting improved health outcomes. Lancet. 2015 Apr 27;385 Suppl 2:S11. doi: 10.1016/S0140-6736(15)60806-6. Epub 2015 Apr 26. PMID 26313057
- [Background] Monk TG, Bronsert MR, Henderson WG, Mangione MP, Sum-Ping ST, Bentt DR, Nguyen JD, Richman JS, Meguid RA, Hammermeister KE. Association between Intraoperative Hypotension and Hypertension and 30-day Postoperative Mortality in Noncardiac Surgery. Anesthesiology. 2015 Aug;123(2):307-19. doi: 10.1097/ALN.0000000000000756. PMID 26083768
- [Background] Sessler DI, Meyhoff CS, Zimmerman NM, Mao G, Leslie K, Vasquez SM, Balaji P, Alvarez-Garcia J, Cavalcanti AB, Parlow JL, Rahate PV, Seeberger MD, Gossetti B, Walker SA, Premchand RK, Dahl RM, Duceppe E, Rodseth R, Botto F, Devereaux PJ. Period-dependent Associations between Hypotension during and for Four Days after Noncardiac Surgery and a Composite of Myocardial Infarction and Death: A Substudy of the POISE-2 Trial. Anesthesiology. 2018 Feb;128(2):317-327. doi: 10.1097/ALN.0000000000001985. PMID 29189290
- [Background] Walsh M, Devereaux PJ, Garg AX, Kurz A, Turan A, Rodseth RN, Cywinski J, Thabane L, Sessler DI. Relationship between intraoperative mean arterial pressure and clinical outcomes after noncardiac surgery: toward an empirical definition of hypotension. Anesthesiology. 2013 Sep;119(3):507-15. doi: 10.1097/ALN.0b013e3182a10e26. PMID 23835589
- [Background] Sun LY, Wijeysundera DN, Tait GA, Beattie WS. Association of intraoperative hypotension with acute kidney injury after elective noncardiac surgery. Anesthesiology. 2015 Sep;123(3):515-23. doi: 10.1097/ALN.0000000000000765. PMID 26181335
- [Background] Wesselink EM, Kappen TH, Torn HM, Slooter AJC, van Klei WA. Intraoperative hypotension and the risk of postoperative adverse outcomes: a systematic review. Br J Anaesth. 2018 Oct;121(4):706-721. doi: 10.1016/j.bja.2018.04.036. Epub 2018 Jun 20. PMID 30236233
- [Background] Futier E, Lefrant JY, Guinot PG, Godet T, Lorne E, Cuvillon P, Bertran S, Leone M, Pastene B, Piriou V, Molliex S, Albanese J, Julia JM, Tavernier B, Imhoff E, Bazin JE, Constantin JM, Pereira B, Jaber S; INPRESS Study Group. Effect of Individualized vs Standard Blood Pressure Management Strategies on Postoperative Organ Dysfunction Among High-Risk Patients Undergoing Major Surgery: A Randomized Clinical Trial. JAMA. 2017 Oct 10;318(14):1346-1357. doi: 10.1001/jama.2017.14172. PMID 28973220
- [Background] Memis D, Hekimoglu S, Vatan I, Yandim T, Yuksel M, Sut N. Effects of midazolam and dexmedetomidine on inflammatory responses and gastric intramucosal pH to sepsis, in critically ill patients. Br J Anaesth. 2007 Apr;98(4):550-2. doi: 10.1093/bja/aem017. No abstract available. PMID 17363413
- [Background] Xiang H, Hu B, Li Z, Li J. Dexmedetomidine controls systemic cytokine levels through the cholinergic anti-inflammatory pathway. Inflammation. 2014 Oct;37(5):1763-70. doi: 10.1007/s10753-014-9906-1. PMID 24803295
- [Background] Cho JS, Kim HI, Lee KY, An JY, Bai SJ, Cho JY, Yoo YC. Effect of Intraoperative Dexmedetomidine Infusion on Postoperative Bowel Movements in Patients Undergoing Laparoscopic Gastrectomy: A Prospective, Randomized, Placebo-Controlled Study. Medicine (Baltimore). 2015 Jun;94(24):e959. doi: 10.1097/MD.0000000000000959. PMID 26091461
- [Background] Kocoglu H, Karaaslan K, Gonca E, Bozdogan O, Gulcu N. Preconditionin effects of dexmedetomidine on myocardial ischemia/reperfusion injury in rats. Curr Ther Res Clin Exp. 2008 Apr;69(2):150-8. doi: 10.1016/j.curtheres.2008.04.003. PMID 24692794
- [Background] Cheng J, Zhu P, Qin H, Li X, Yu H, Yu H, Peng X. Dexmedetomidine attenuates cerebral ischemia/reperfusion injury in neonatal rats by inhibiting TLR4 signaling. J Int Med Res. 2018 Jul;46(7):2925-2932. doi: 10.1177/0300060518781382. Epub 2018 Jun 21. PMID 29926753
- [Background] Sahin T, Begec Z, Toprak HI, Polat A, Vardi N, Yucel A, Durmus M, Ersoy MO. The effects of dexmedetomidine on liver ischemia-reperfusion injury in rats. J Surg Res. 2013 Jul;183(1):385-90. doi: 10.1016/j.jss.2012.11.034. Epub 2012 Dec 8. PMID 23321519
- [Background] Hanci V, Yurdakan G, Yurtlu S, Turan IO, Sipahi EY. Protective effect of dexmedetomidine in a rat model of alpha-naphthylthiourea-induced acute lung injury. J Surg Res. 2012 Nov;178(1):424-30. doi: 10.1016/j.jss.2012.02.027. Epub 2012 Mar 9. PMID 22445456
- [Background] Kocoglu H, Ozturk H, Ozturk H, Yilmaz F, Gulcu N. Effect of dexmedetomidine on ischemia-reperfusion injury in rat kidney: a histopathologic study. Ren Fail. 2009;31(1):70-4. doi: 10.1080/08860220802546487. PMID 19142813
- [Background] Duncan D, Sankar A, Beattie WS, Wijeysundera DN. Alpha-2 adrenergic agonists for the prevention of cardiac complications among adults undergoing surgery. Cochrane Database Syst Rev. 2018 Mar 6;3(3):CD004126. doi: 10.1002/14651858.CD004126.pub3. PMID 29509957
- [Background] Kheterpal S, Tremper KK, Heung M, Rosenberg AL, Englesbe M, Shanks AM, Campbell DA Jr. Development and validation of an acute kidney injury risk index for patients undergoing general surgery: results from a national data set. Anesthesiology. 2009 Mar;110(3):505-15. doi: 10.1097/ALN.0b013e3181979440. PMID 19212261
- [Background] Marik PE, Cavallazzi R, Vasu T, Hirani A. Dynamic changes in arterial waveform derived variables and fluid responsiveness in mechanically ventilated patients: a systematic review of the literature. Crit Care Med. 2009 Sep;37(9):2642-7. doi: 10.1097/CCM.0b013e3181a590da. PMID 19602972
- [Background] Khwannimit B, Bhurayanontachai R. Prediction of fluid responsiveness in septic shock patients: comparing stroke volume variation by FloTrac/Vigileo and automated pulse pressure variation. Eur J Anaesthesiol. 2012 Feb;29(2):64-9. doi: 10.1097/EJA.0b013e32834b7d82. PMID 21946822
- [Background] Trepte CJ, Eichhorn V, Haas SA, Stahl K, Schmid F, Nitzschke R, Goetz AE, Reuter DA. Comparison of an automated respiratory systolic variation test with dynamic preload indicators to predict fluid responsiveness after major surgery. Br J Anaesth. 2013 Nov;111(5):736-42. doi: 10.1093/bja/aet204. Epub 2013 Jun 27. PMID 23811425
- [Background] Katayama H, Kurokawa Y, Nakamura K, Ito H, Kanemitsu Y, Masuda N, Tsubosa Y, Satoh T, Yokomizo A, Fukuda H, Sasako M. Extended Clavien-Dindo classification of surgical complications: Japan Clinical Oncology Group postoperative complications criteria. Surg Today. 2016 Jun;46(6):668-85. doi: 10.1007/s00595-015-1236-x. Epub 2015 Aug 20. PMID 26289837
- [Background] Kellum JA, Lameire N; KDIGO AKI Guideline Work Group. Diagnosis, evaluation, and management of acute kidney injury: a KDIGO summary (Part 1). Crit Care. 2013 Feb 4;17(1):204. doi: 10.1186/cc11454. PMID 23394211
- [Background] Yang L, Xing G, Wang L, Wu Y, Li S, Xu G, He Q, Chen J, Chen M, Liu X, Zhu Z, Yang L, Lian X, Ding F, Li Y, Wang H, Wang J, Wang R, Mei C, Xu J, Li R, Cao J, Zhang L, Wang Y, Xu J, Bao B, Liu B, Chen H, Li S, Zha Y, Luo Q, Chen D, Shen Y, Liao Y, Zhang Z, Wang X, Zhang K, Liu L, Mao P, Guo C, Li J, Wang Z, Bai S, Shi S, Wang Y, Wang J, Liu Z, Wang F, Huang D, Wang S, Ge S, Shen Q, Zhang P, Wu L, Pan M, Zou X, Zhu P, Zhao J, Zhou M, Yang L, Hu W, Wang J, Liu B, Zhang T, Han J, Wen T, Zhao M, Wang H; ISN AKF 0by25 China Consortiums. Acute kidney injury in China: a cross-sectional survey. Lancet. 2015 Oct 10;386(10002):1465-71. doi: 10.1016/S0140-6736(15)00344-X. PMID 26466051
- [Background] Fourth universal definition of myocardial infarction (2018). Rev Esp Cardiol (Engl Ed). 2019 Jan;72(1):72. doi: 10.1016/j.rec.2018.11.011. No abstract available. English, Spanish. PMID 30580786
- [Background] Canet J, Gallart L, Gomar C, Paluzie G, Valles J, Castillo J, Sabate S, Mazo V, Briones Z, Sanchis J; ARISCAT Group. Prediction of postoperative pulmonary complications in a population-based surgical cohort. Anesthesiology. 2010 Dec;113(6):1338-50. doi: 10.1097/ALN.0b013e3181fc6e0a. PMID 21045639
- [Background] Bernard GR, Artigas A, Brigham KL, Carlet J, Falke K, Hudson L, Lamy M, Legall JR, Morris A, Spragg R. The American-European Consensus Conference on ARDS. Definitions, mechanisms, relevant outcomes, and clinical trial coordination. Am J Respir Crit Care Med. 1994 Mar;149(3 Pt 1):818-24. doi: 10.1164/ajrccm.149.3.7509706.
- [Background] Easton JD, Saver JL, Albers GW, Alberts MJ, Chaturvedi S, Feldmann E, Hatsukami TS, Higashida RT, Johnston SC, Kidwell CS, Lutsep HL, Miller E, Sacco RL; American Heart Association; American Stroke Association Stroke Council; Council on Cardiovascular Surgery and Anesthesia; Council on Cardiovascular Radiology and Intervention; Council on Cardiovascular Nursing; Interdisciplinary Council on Peripheral Vascular Disease. Definition and evaluation of transient ischemic attack: a scientific statement for healthcare professionals from the American Heart Association/American Stroke Association Stroke Council; Council on Cardiovascular Surgery and Anesthesia; Council on Cardiovascular Radiology and Intervention; Council on Cardiovascular Nursing; and the Interdisciplinary Council on Peripheral Vascular Disease. The American Academy of Neurology affirms the value of this statement as an educational tool for neurologists. Stroke. 2009 Jun;40(6):2276-93. doi: 10.1161/STROKEAHA.108.192218. Epub 2009 May 7. PMID 19423857
- [Background] Ely EW, Margolin R, Francis J, May L, Truman B, Dittus R, Speroff T, Gautam S, Bernard GR, Inouye SK. Evaluation of delirium in critically ill patients: validation of the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU). Crit Care Med. 2001 Jul;29(7):1370-9. doi: 10.1097/00003246-200107000-00012. PMID 11445689
- [Background] Konstantinides SV. 2014 ESC Guidelines on the diagnosis and management of acute pulmonary embolism. Eur Heart J. 2014 Dec 1;35(45):3145-6. doi: 10.1093/eurheartj/ehu393. No abstract available. PMID 25452462
- [Background] Scarvelis D, Wells PS. Diagnosis and treatment of deep-vein thrombosis. CMAJ. 2006 Oct 24;175(9):1087-92. doi: 10.1503/cmaj.060366. PMID 17060659
- [Background] Horan TC, Andrus M, Dudeck MA. CDC/NHSN surveillance definition of health care-associated infection and criteria for specific types of infections in the acute care setting. Am J Infect Control. 2008 Jun;36(5):309-32. doi: 10.1016/j.ajic.2008.03.002. No abstract available. PMID 18538699
- [Background] Seymour CW, Liu VX, Iwashyna TJ, Brunkhorst FM, Rea TD, Scherag A, Rubenfeld G, Kahn JM, Shankar-Hari M, Singer M, Deutschman CS, Escobar GJ, Angus DC. Assessment of Clinical Criteria for Sepsis: For the Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):762-74. doi: 10.1001/jama.2016.0288. PMID 26903335